CLINICAL TRIAL: NCT04320589
Title: The Perioperative Use of Dexmedetomidine and Magnesium Sulfate Compared With Traditional Anesthetic Technique for Open Resection of Pheochromocytoma.
Brief Title: the Effect of Dexmedetomidine and Magnesium Sulfate in Open Resection of Pheochromocytoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ehab Hanafy Shaker, lecturer of anesthesia ,critical care and pain medicine, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ehab - Hegazy pheochromocytoma
Record Dates: First submitted 2020-03-22; First posted 2020-03-25 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Pheochromocytoma
MeSH Terms: conditions — Pheochromocytoma | interventions — Dexmedetomidine; Anesthetics, General; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Active Comparator): Traditional group in which the patients̕ hemodynamic adjustment will be conducted using orally or IV α₁ & β-adrenergic blockers [Prazosin (minipress): 0.5-20 mg/day, Propranolol (Inderal) :10-360 mg/day, Bisoprolol (Concor): 2.5-20 mg/day, Atenolol (Tenormin): 25-100 mg/day &/or Labetalol (Trandate)200-600 mg/day, Angiotensin Converting enzyme inhibitors ( ACE inhibitors ) & Angiotensin II receptor blockers ARBs e.g. Tritace 2.5-10 mg/day & Atacand 4-16 mg/day]
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine (Active Comparator): Dexmedetomidine-Magnesium Sulfate (Dex-MgSo₄) group: in which in addition to the orally prescribed drugs; on admission to the ICU, the Pheo-patient has serum-Mg level measurement & a bolus of 40 mg/kg MgSo₄ is given I.V. & may be repeated until the therapeutic level of MgSo₄ 2-4 mmol/Liter is reached. Dexmedetomidine sedation is started the evening prior to surgery by loading dose of 1µg/Kg followed by 0.2-0.7 µg/Kg/hour according to each patient
  Interventions: Drug: General anesthetic

INTERVENTIONS:
Drug: Dexmedetomidine — which in addition to the orally prescribed drugs; on admission to the ICU, the Pheo-patient has serum-Mg level measurement & a bolus of 40 mg/kg MgSo₄ is given I.V. & may be repeated until the therapeutic level of MgSo₄ 2-4 mmol/Liter is reached (7&10). Dexmedetomidine sedation is started the evening prior to surgery by loading dose of 1µg/Kg followed by 0.2-0.7 µg/Kg/hour according to each patient
  Other Names: drug group
  Arms: General Anesthesia
Drug: General anesthetic — 1) Traditional group in which the patients̕ hemodynamic adjustment will be conducted using orally or IV α₁ & β-adrenergic blockers [Prazocin (minipress): 0.5-20 mg/day, Propranolol (Inderal) :10-360 mg/day, Bisoprolol (Concor): 2.5-20 mg/day, Atenolol (Tenormin): 25-100 mg/day &/or Labetalol (Trandate)200-600 mg/day, ACI & ACRB e.g. Tritace 2.5-10 mg/day & Atacand 4-16 mg/day]
  Other Names: control group
  Arms: Dexmedetomidine

SUMMARY:
Pheochromocytoma (pheo) is a catecholamine secreting tumor arising from chromaffin cells of the adrenal medulla in 90% of cases & in 10% is extra-adrenal arising from the sympathetic chain. It is malignant in 10% of cases, bilateral in 10% of patients & 10% of all pheo are inherited (Familial Pheo) as autosomal dominant either alone or as a part of multiple endocrine neoplasia (MEN) syndrome.In this prospective work, the investigators will try to compare the peri-operative hemodynamic course of Dexmedetomidine & magnesium sulphate (MgSo₄) infused patients with the traditional anesthetic technique (α₁ & β-adrenergic blockers plus vasodilators) during open surgical resection of Pheo. The investigators are aiming to check the safety & efficacy of the recommended technique on the peri-operative hemodynamic stability & controlling the hypertensive crisis during tumor manipulation.

DETAILED DESCRIPTION:
Pheochromocytoma (pheo) is a catecholamine secreting tumor arising from chromaffin cells of the adrenal medulla in 90% of cases & in 10% is extra-adrenal arising from the sympathetic chain. It is malignant in 10% of cases, bilateral in 10% of patients & 10% of all pheo are inherited (Familial Pheo) as autosomal dominant either alone or as a part of multiple endocrine neoplasia (MEN) syndrome.The anesthetic management of Pheo during surgical resection is usually challenging & faces many cardiovascular risks as tachycardia, arrhythmias, severe hypertension & may be pulmonary edema & profound hypotension after surgical devascularization of the tumor. These dangerous events are sequelae of catecholamine excess and often are refractory to management . The proper anesthetic control is based on the use of α₁ & β-adrenergic blockers (phenoxy-benzamine, phentolamine, propranolol, labetalol) and vasodilators such as glycerine trinitrate (GTN) & sodium nitroprusside (SNP) .The rational of using magnesium sulphate MgSo₄ infusion to control catecholamine levels & catecholamine-related crisis has been established in several clinical emergencies such as severe tetanus & preoperative management of pre-eclampsia & eclampsia . MgSo₄ beneficial cardiovascular effects may be attributed to its ability to reduce catecholamine release from the adrenal medulla & to reduce α-adrenergic receptors sensitivity to catecholamines . MgSo₄ is also a direct vasodilator & a potent anti-arrhythmic drug particularly with high circulatory catecholamine level . The safety of MgSo₄ in the routine clinical range of 2-4 mmol/Liter is well settled in many clinical works.

There is strong evidence that the sympathetic nervous system is intact in Pheo patients & neurons-released noradrenaline plays a fundamental role in blood pressure BP regulation. Dexmedetomidine is a short acting & highly selective central α₂-agonist that inhibits neuronal firing & thereby induces analgesia, anxiolysis, bradycardia & hypotension. It has been tried to attenuate the sympathetic pressor effect of tracheal intubation, cardiac surgeries & emergence from anesthesia .The unique adventitious anesthetic pharmacology induces preoperative sedation, intra-operative hemodynamic stability beside reducing the anesthetic requirements and adding to post-operative analgesia . Its peri-operative use has been suggested in both pediatric & adult patients of Pheo.

In this prospective work,the investigators tried to compare the peri-operative hemodynamic course of Dexmedetomidine & MgSo₄ infused patients with the traditional anesthetic technique (α₁ & β-adrenergic blockers plus vasodilators) during open surgical resection of Pheo. The investigators are aiming to check the safety & efficacy of this recommended technique on the peri-operative hemodynamic stability & controlling the hypertensive crisis during tumor manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-69 years
* ASA physical status I &II
* Surgically diagnosed pheochromocytoma, "unilateral or bilateral, adrenal or extra-adrenal". Diagnosis is confirmed radiologically with or without laboratory Vanillyl Mandelic Acid (VMA) level.
* Accepted Echo-heart data (EF ≥ 55%, no serious valve lesion) apart from hypertensive concentric ventricular hypertrophy & diastolic dysfunction grade I &II.

Exclusion Criteria:

* Extremes of age
* ASA III & IV
* History of cardiac (MI & IHD) or cerebral (CVS) events
* History of major reaction to the used drugs
* History of major muscle, endocrinal or hematologic disorders
* Pregnant and lactating women
* Poor Echo-heart findings e.g. EF < 55%, severe valve lesions & severe pulmonary hypertension.

Ages: 12 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
The rate of Hypertensive crisis | 12 hours follow up
  rise of B.P. more than 20% of base line

CONTACTS AND LOCATIONS:
Overall Officials: Ehab H Shaker, MD, Principal Investigator — National Cancer Institute- Cairo University
Locations (1):
- Department of Anesthesia and Pain medicine.National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
After total completion of the study

REFERENCES:
- See also: Dexmedetomidine as intravenous sedating agent — https://anesthesiology.pubs.asahq.org/article.aspx?articleid=1942849